CLINICAL TRIAL: NCT04629729
Title: A Phase I Study of FT819 in Subjects With B-cell Malignancies
Brief Title: FT819 in Subjects With B-cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT819-101
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, B-Cell; Chronic Lymphocytic Leukemia; Precursor B-Cell Acute Lymphoblastic Leukemia
Keywords: Lymphoma; Leukemia; BCL; CLL; B-ALL; CAR-T; cellular therapy
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Leukemia | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- FT819 Single-Dose Monotherapy, B-Cell Lymphoma (Experimental): FT819 single-dose monotherapy in adult subjects with r/r B-cell Lymphoma
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT819 Single-Dose in Combination with IL-2, B-Cell Lymphoma (Experimental): FT819 single-dose in combination with IL-2 in adult subjects with r/r B-cell Lymphoma
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2; Drug: Bendamustine
- FT819 Step Fractionated Monotherapy, B-Cell Lymphoma (Experimental): FT819 monotherapy administered as step-fractionated dosing in adult subjects with r/r B-cell Lymphoma
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT819 Single-Dose Monotherapy, CLL (Experimental): FT819 single-dose monotherapy in adult subjects with r/r CLL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT819 Single-Dose in Combination with IL-2, CLL (Experimental): FT819 single-dose in combination with IL-2 in adult subjects with r/r CLL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2; Drug: Bendamustine
- FT819 Step Fractionated Monotherapy, CLL (Experimental): FT819 monotherapy administered as step-fractionated dosing in adult subjects with r/r CLL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT819 Single-Dose Monotherapy, B-ALL (Experimental): FT819 single-dose monotherapy in adult subjects with r/r B-ALL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT819 Single-Dose in Combination with IL-2, B-ALL (Experimental): FT819 single-dose in combination with IL-2 in adult subjects with r/r B-ALL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2; Drug: Bendamustine
- FT819 Step Fractionated Monotherapy, B-ALL (Experimental): FT819 monotherapy administered as step-fractionated dosing in adult subjects with r/r B-ALL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- FT819 Step Fractionated Monotherapy in Combination with IL-2, B-Cell Lymphoma (Experimental): FT819 monotherapy administered as step-fractionated dosing in combination with IL-2 in adult subjects with r/r B-cell Lymphoma
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2; Drug: Bendamustine
- FT819 Step Fractionated Monotherapy in Combination with IL-2, CLL (Experimental): FT819 monotherapy administered as step-fractionated dosing in combination with IL-2 in adult subjects with r/r CLL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2; Drug: Bendamustine
- FT819 Step Fractionated Monotherapy in Combination with IL-2, B-ALL (Experimental): FT819 monotherapy administered as step-fractionated dosing in combination with IL-2 in adult subjects with r/r B-ALL
  Interventions: Drug: FT819; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2; Drug: Bendamustine

INTERVENTIONS:
Drug: FT819 — Experimental Interventional Therapy
Drug: Cyclophosphamide — Lympho-conditioning agent
Drug: Fludarabine — Lympho-conditioning agent
  Other Names: Fludara
Drug: IL-2 — Biologic response modifier
  Other Names: Interleukin-2
  Arms: FT819 Single-Dose in Combination with IL-2, B-ALL; FT819 Single-Dose in Combination with IL-2, B-Cell Lymphoma; FT819 Single-Dose in Combination with IL-2, CLL; FT819 Step Fractionated Monotherapy in Combination with IL-2, B-ALL; FT819 Step Fractionated Monotherapy in Combination with IL-2, B-Cell Lymphoma; FT819 Step Fractionated Monotherapy in Combination with IL-2, CLL
Drug: Bendamustine — Lympho-conditioning agent
  Other Names: Bendeka; Treanda

SUMMARY:
This is a Phase I dose-finding study of FT819 as monotherapy and in combination with IL-2 in subjects with relapsed/refractory B-cell Lymphoma, Chronic Lymphocytic Leukemia and Precursor B-cell Acute Lymphoblastic Leukemia. The study will consist of a dose-escalation stage and an expansion stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

Diagnosis of B-cell lymphoma, CLL or B-ALL as described below:

B-Cell Lymphoma:

* Histologically documented lymphomas expected to express CD19
* Relapsed/refractory disease following at least 2 prior lines of multi-agent immunochemotherapy

Chronic Lymphocytic Leukemia (CLL):

* Diagnosis of CLL per iwCLL guidelines
* Relapsed/refractory disease following at least two prior systemic treatment regimens

Precursor B-cell Acute Lymphocytic Leukemia (B-ALL):

* Diagnosis of B-ALL by flow cytometry, bone marrow histology, and/or cytogenetics
* Relapsed/refractory disease after at least 2 cycles of standard multiagent induction chemotherapy. For subjects with Philadelphia-chromosome positive (Ph+) disease, failure or intolerance to a tyrosine kinase inhibitor therapy-containing regimen

ALL SUBJECTS:

* Capable of giving signed informed consent
* Age ≥ 18 years old
* Stated willingness to comply with study procedures and duration
* Contraceptive use for women and men as defined in the protocol

Key Exclusion Criteria:

ALL SUBJECTS:

* Females who are pregnant or breastfeeding
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥2
* Body weight <50 kg
* Evidence of insufficient organ function
* Receipt of therapy within 2 weeks prior to Day 1 or five half-lives, whichever is shorter; or any investigational therapy within 28 days prior to Day 1
* Currently receiving or likely to require systemic immunosuppressive therapy
* Ongoing requirement for systemic GvHD therapy following prior allogeneic hematopoietic stem cell transplant (HSCT) or allogeneic CAR-T
* Receipt of an allograft organ transplant
* Known active central nervous system (CNS) involvement by malignancy
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Clinically significant cardiovascular disease
* Positive serologic test results for HIV infection
* Positive serologic and polymerase chain reaction (PCR) test results for Hepatitis B (HBV) infection
* Positive serologic and PCR test results for Hepatitis C (HCV) infection
* Live vaccine <6 weeks prior to start of lympho-conditioning
* Known allergy to albumin (human) or DMSO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2039-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities within each dose level cohort | Up to Day 29
Incidence, nature, and severity of adverse events (AEs) of FT819 as monotherapy and in combination with IL-2 in r/r B-cell lymphoma, r/r chronic lymphocytic leukemia, and r/r precursor B-cell acute lymphoblastic leukemia | Up to 15 years

SECONDARY OUTCOMES:
Investigator-assessed objective-response rate (ORR) | Up to approximately 2 years after last dose of FT819
For BCL and CLL Only: Investigator-assessed duration of objective response (DOR) | Up to 15 years
For BCL and CLL Only: Investigator-assessed duration of complete response (DoCR) | Up to 15 years
For BCL and CLL Only: Progression-free survival (PFS) | Up to 15 years
Overall survival (OS) | Up to 15 years
Determination of the pharmacokinetics of FT819 cells in peripheral blood. | Study Days 1, 2, 3, 4, 5, 8, 11, 15, 22, and 29
  The PK of FT819 in peripheral blood will be reported as the relative percentage of product (FT819) DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points
For B-ALL Only: Investigator-assessed relapse-free survival (RFS) | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Arizona, Phoenix, Arizona
  - UC Davis, Davis, California
  - Scripps Green Hospital, La Jolla, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Mayo Florida, Jacksonville, Florida
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Mayo Minnesota, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Sciences University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ASH 2022 Poster Presentation — https://fatetherapeutics.com/wp-content/uploads/2022/12/2000-FT81989.pdf
- See also: ASH 2022 Abstract — https://ash.confex.com/ash/2022/webprogram/Paper167194.html